CLINICAL TRIAL: NCT00682565
Title: Tolerability and CK-1827452 Plasma Concentrations During Intravenous and Immediate-Release Oral CK-1827452 in Patients With Ischemic Cardiomyopathy and Angina
Brief Title: PK and Tolerability of IV and Oral CK-1827452 in Patients With Ischemic Cardiomyopathy and Angina
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 1221
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Results first posted 2010-02-25 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2010-02

CONDITIONS: Heart Failure; Myocardial Ischemia; Angina Pectoris
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia; Angina Pectoris | interventions — omecamtiv mecarbil; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Mid Dose CK-1827452 or Placebo (Experimental): CK-1827452 I.V. infusion for 2 hours at 24mg/hr followed by 18 hours at 6mg/hr or placebo, followed by 6 days three times a day oral dose and a final single oral dose
  Interventions: Drug: CK-1827452 24mg and 6 mg iv infusion; Drug: CK-1827452 12.5mg capsule; Drug: Placebo iv infusion; Drug: Placebo capsule
- High Dose CK-1827452 or Placebo (Experimental): CK-1827452 I.V. infusion for 2 hours at 48mg/hr followed by 18 hours at 11mg/hr or placebo, followed by 6 days three times a day oral dose and a final single oral dose
  Interventions: Drug: CK-1827452 48 mg and 11 mg iv infusion; Drug: CK-1827452 25mg capsule; Drug: Placebo iv infusion; Drug: Placebo capsule

INTERVENTIONS:
Drug: CK-1827452 24mg and 6 mg iv infusion — I.V. infusion for 2 hours at 24mg/hr followed by 18 hours at 6mg/hr
  Other Names: omecamtiv mecarbil
  Arms: Mid Dose CK-1827452 or Placebo
Drug: CK-1827452 12.5mg capsule — 12.5mg oral immediate release capsule
  Other Names: omecamtiv mecarbil
  Arms: Mid Dose CK-1827452 or Placebo
Drug: CK-1827452 48 mg and 11 mg iv infusion — I.V. infusion for 2 hours at 48mg/hr followed by 18 hours at 11mg/hr
  Other Names: omecamtiv mecarbil
  Arms: High Dose CK-1827452 or Placebo
Drug: CK-1827452 25mg capsule — 25mg oral immediate release capsule
  Other Names: omecamtiv mecarbil
  Arms: High Dose CK-1827452 or Placebo
Drug: Placebo iv infusion — Matching placebo iv infusion
Drug: Placebo capsule — Matching placebo oral immediate release capsule

SUMMARY:
This study investigates whether symptom-limited exercise capacity in ischemic cardiomyopathy patients with angina is deleteriously affected by treatment with CK-1827452.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effect of intravenous (i.v.) CK-1827452 on symptom-limited exercise tolerance in patients with ischemic cardiomyopathy and angina. The secondary objectives are to assess the tolerability of CK-1827452 administered three times daily (tid) to steady state in an immediate-release (IR), blend-in-capsule oral formulation to outpatients with ischemic cardiomyopathy and angina and to assess CK-1827452 plasma concentrations at trough and 1 hour after dosing with CK-1827452 administered tid to steady state in an IR, blend-in-capsule oral formulation to outpatients with ischemic cardiomyopathy and angina.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed an Informed Consent Form/Patient Information Sheet for this study approved by the governing Institutional Review Board (IRB) or Independent Ethics Committee (IEC).
2. The patient is at least 18 years old.
3. The patient has ischemic heart disease documented by any one or more of the following:

   * A history of myocardial infarction documented by elevated CPK-MB, troponin I or T, or the presence of electrocardiographic Q waves consistent with myocardial infarction.
   * Coronary angiography demonstrating at least 1 major epicardial coronary artery (i.e., left main, left anterior descending, left circumflex, or right coronary artery) with a stenosis of at least 60% diameter or greater but excluding stenosis of the left main coronary artery unless revascularized by coronary artery bypass grafting.
4. The patient has a history of ≥ 1 episode of exercise induced angina within 2 months prior to the initial screening visit.
5. The patient has been taking a beta blocker and an ACE inhibitor (and/or an ARB) for at least 4 weeks. If prescribed, diuretics must have been administered for at least 4 weeks prior to the initial screening visit.
6. The patient is NYHA Class II-III at the time of enrollment and has been so for ≥ 3 months prior to the initial screening visit.
7. The patient has a history of a left ventricular ejection fraction (LVEF) ≤ 35%.
8. The patient has a history of EITHER a left ventricular end-diastolic diameter ≥ 55 mm, OR a left ventricular end-diastolic diameter index ≥ 32 mm/m2.
9. The patient can be expected to complete at least 4 minutes of a Modified Naughton ETT (see Appendix B).
10. For female patients only: The patient is post-menopausal (≥ 1 year) or sterilized, or if she is of childbearing potential, she is not breastfeeding, her pregnancy test is negative, she has no intention to become pregnant during the course of the study, and she is using contraceptive drugs or devices.

Exclusion Criteria:

1. The patient has acute myocarditis; clinically significant restrictive, constrictive, or hypertrophic obstructive cardiomyopathy; or clinically significant congenital heart disease.
2. The patient has a SBP > 160 mmHg, documented on at least 3 separate occasions, at least 10 minutes apart.
3. The patient has a DBP > 90 mmHg, documented on at least 3 separate occasions, at least 10 minutes apart.
4. The patient has levels of troponin I or T, or CPK-MB > the upper limit of normal at any time from 6 weeks prior to the Initial Screening Visit (Visit 1) and up to randomization.
5. The patient has severe aortic or mitral stenosis.
6. The patient has had an acute coronary syndrome, transient ischemic attack, or revascularization procedure within 6 weeks of the Initial Screening Visit (Visit 1).
7. The patient has significant co-morbid conditions (i.e., lung disease, arthritis, peripheral vascular disease) that may limit his or her treadmill exercise capacity.
8. The patient has renal impairment defined by a calculated creatinine clearance < 30 cc/min or a need for renal replacement therapy.
9. The patient has known hepatic impairment defined by a total bilirubin > 3 mg/dL, or an ALT or AST > 2 times the upper limit of normal.
10. The patient has received an investigational drug or device within 30 days or 5 half-lives, whichever is greater, of randomization.
11. The patient weighs > 120 kg.
12. The patient has a body temperature > 38 ° C, confirmed by at least 2 successive measurements, at least 10 minutes apart.
13. The patient has any laboratory abnormality which, in the opinion of the investigator, should preclude his or her participation in the study.
14. The patient has had any prior treatment with CK-1827452.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Wolff, MD, FACC, Study Chair — Cytokinetics, Inc.
Locations (14):
- Georgia (6):
  - Tbilisi State Medical University Clinic #1, Tbilisi
  - Cardio-Reanimation Centre, Tbilisi
  - Cardiology Clinic, Tbilisi
  - National Center of Therapy, Tbilisi
  - Multiprofile Clinical Hospital of Tbilisi #2, Tbilisi
  - Diagnostic Services Clinic, Tbilisi
- Russia (8):
  - Altay Territory Cardiology Dispensary, Barnaul
  - City Hospital #1, Barnaul
  - City Clinical Hospital #59, Moscow
  - City Clinical Hospital #64, Moscow
  - Moscow Municipal Clinical Hospital #4, Moscow
  - Federal Center of Heart, Blood and Endocrinology n.a. Almazov, Saint Petersburg
  - Research Centre for Cardiology n.a. Almazov under Roszdrav, Saint Petersburg
  - Volgograd Regional Cardiology Center, Volgograd

REFERENCES:
- [Derived] Greenberg BH, Chou W, Saikali KG, Escandon R, Lee JH, Chen MM, Treshkur T, Megreladze I, Wasserman SM, Eisenberg P, Malik FI, Wolff AA, Shaburishvili T. Safety and tolerability of omecamtiv mecarbil during exercise in patients with ischemic cardiomyopathy and angina. JACC Heart Fail. 2015 Jan;3(1):22-29. doi: 10.1016/j.jchf.2014.07.009. Epub 2014 Nov 11. PMID 25453536

RESULTS

PARTICIPANT FLOW:
Groups:
- Mid Dose CK-1827452; High Dose CK-1827452: CK-1827452 20 hour infusion followed by 6 days three times a day oral dose and a final single oral dose
- Placebo: 20 hour infusion followed by 6 days three times a day oral dose and a final single oral dose
Period: Overall Study
Arm/Group | Mid Dose CK-1827452 | High Dose CK-1827452 | Placebo
Started | 31 | 35 | 29
Completed | 30 | 32 | 29
Not Completed | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mid Dose Active Drug; High Dose Active Drug: CK-1827452 20 hour infusion followed by 6 days three times a day oral dose and a final single oral dose
- All Placebo: 20 hour infusion followed by 6 days three times a day oral dose and a final single oral dose
- Total: Total of all reporting groups
Arm/Group | Mid Dose Active Drug | High Dose Active Drug | All Placebo | Total
Number analyzed (Participants) | 31 | 34 | 29 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 16 | 17 | 44
  >=65 years | 20 | 18 | 12 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.0) | 62.6 (8.1) | 62.3 (9.8) | 63.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 6 | 19
  Male | 23 | 29 | 23 | 75
Region of Enrollment [Number; unit: participants]
  Russian Federation | 0 | 14 | 7 | 21
  Georgia | 31 | 20 | 22 | 73

OUTCOME MEASURES:

1. Primary Outcome: Participants Stopping Exercise Treadmill Test 3 (ETT-3) for Angina at Stage Earlier Than Baseline Exercise Treadmill Test (ETT-B)
Description: The Modified Naughton Exercise Treadmill Test was employed in this study. Exercise Treadmill Test 3 (ETT-3) was performed during the last 2 hours of the 20-hour infusion of study drug or placebo. Baseline Exercise Treadmill Test (ETT-B) was performed prior to dosing.
Time Frame: 1 day
Population: The Safety ETT Population consists of all patients in the Randomized Population who received any study drug and who performed ETT-3.
Measure: Number; unit: Participants
Arm/Group | Mid Dose Active Drug | High Dose Active Drug | All Placebo
Number analyzed (Participants) | 31 | 34 | 29
Participants | 0 | 0 | 1

2. Secondary Outcome: Participants Stopping ETT-3 for Any Reason at Stage Earlier Than ETT-B
Description: as for outcome 1
Time Frame: 1 day
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Mid Dose Active Drug | High Dose Active Drug | All Placebo
Number analyzed (Participants) | 31 | 34 | 29
Participants | 4 | 2 | 1

3. Secondary Outcome: Increase in Exercise Duration During ETT-3 vs. ETT-B
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Mid Dose Active Drug | High Dose Active Drug | All Placebo
Number analyzed (Participants) | 31 | 34 | 29
seconds | 41.5 (113.1) | 40.5 (70.6) | 60.1 (71.2)

4. Secondary Outcome: Participants Stopping ETT-3 for Angina at Any Stage
Description: This Outcome Measure includes all participants who stopped ETT-3 for angina at any stage, not only those who stopped at a stage earlier than ETT-B.
  Note: All 9 subjects who stopped ETT-3 for angina also stopped ETT-B for angina.
Time Frame: 1 day
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Mid Dose Active Drug | High Dose Active Drug | All Placebo
Number analyzed (Participants) | 31 | 34 | 29
Participants | 0 | 7 | 2

5. Secondary Outcome: Participants With 1 mm ST Segment Depression During ETT-3
Description: ST Segment Depression measured by Electrocardiography while performing ETT-3.
Time Frame: 1 day
Population: The Safety ETT Population consists of all patients in the Randomized Population who received any study drug and who performed ETT-3. However, majority of patients did not have ECGs assessable (per protocol) for 1 mm ST depression.
Measure: Number; unit: Participants
Arm/Group | Mid Dose Active Drug | High Dose Active Drug | All Placebo
Number analyzed (Participants) | 10 | 12 | 7
Participants | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: 2 - 3 weeks
Groups:
- Cohort 1 Active Drug; Cohort 2 Active Drug: CK-1827452 20 hour infusion followed by 6 days three times a day oral dose and a final single oral dose
- Total: All Patients
Arm/Group | Cohort 1 Active Drug | Cohort 2 Active Drug | All Placebo | Total
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/34 | 0/29 | 1/94
Other Adverse Events (participants affected / at risk) | 2/31 | 7/34 | 3/29 | 12/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Active Drug (N=31) | Cohort 2 Active Drug (N=34) | All Placebo (N=29) | Total (N=94)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Reported as unrelated to treatment by Investigator but upgraded to possibly related by the sponsor.
Post-procedural Myocardial Infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Reported as unrelated to treatment by Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Active Drug (N=31) | Cohort 2 Active Drug (N=34) | All Placebo (N=29) | Total (N=94)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Infusion Site Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to publish the results of the trial in collaboration with the Investigators.